CLINICAL TRIAL: NCT03068351
Title: Open-label, Multicenter, Dose-escalation/Expansion Phase Ib Study to Evaluate Safety, Pharmacokinetics, and Activity of BET Inhibitor RO6870810, Given as Mono- and Combination Therapy to Patients With Advanced Multiple Myeloma
Brief Title: Study of Bromodomain and Extra-Terminal Protein (BET) Inhibitor RO6870810 as Mono- and Combination Therapy in Advanced Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP39403; 2016-003615-35 (EudraCT Number)
Record Dates: First submitted 2017-02-27; First posted 2017-03-01 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — RO6870810; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RO6870810 (Experimental): Participants will be administered RO6870810 monotherapy at ascending-dose levels during the dose escalation phase followed by an expansion phase during which RO6870810 will be administered as monotherapy at the recommended dose. Participants will continue to receive study drug as long as they experience clinical benefit in the opinion of the Investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression, as determined by the Investigator after an integrated assessment of IMWG response criteria, biopsies/aspirate (if applicable), and clinical status, or withdrawal of consent.
  Interventions: Drug: RO6870810
- RO6870810 + Daratumumab (Experimental): Participants will be administered RO6870810 at ascending-dose levels in combination with daratumumab at the recommended dose during the dose escalation phase followed by an expansion phase during which both RO6870810 and daratumumab will be administered each at their recommended dose. Participants will continue to receive the study drugs as long as they experience clinical benefit in the opinion of the Investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression, as determined by the Investigator after an integrated assessment of IMWG response criteria, biopsies/aspirate (if applicable), and clinical status, or withdrawal of consent.
  Interventions: Drug: RO6870810; Biological: daratumumab

INTERVENTIONS:
Drug: RO6870810 — RO6870810 will be administered subcutaneously (SC) at ascending-dose levels (from 0.30 milligrams/kilogram [mg/kg] to 0.65 mg/kg). In Cycle 1, RO6870810 will be given on Day 1 (omitted on Day 2) and then every day from Day 3 through to Day 15. Starting at Cycle 2, it will be given every day from Day 1 to Day 14 of each 21-day cycle. In the first combination therapy cohort RO6870810 will be administered at one dose-level below the maximum tolerated dose (MTD).
Biological: daratumumab — Daratumumab will be administered intravenously (IV) at a dose of 16 milligrams/kilogram (mg/kg) of body weight weekly for the first 8 weeks, every two weeks for the following 16 weeks, and every four weeks thereafter, until disease progression.
  Arms: RO6870810 + Daratumumab

SUMMARY:
This is a Phase Ib, open-label, multicenter, global study designed to assess the safety and tolerability of RO6870810 as monotherapy and in combination with daratumumab in participants with relapsed/refractory multiple myeloma. Each treatment cycle will be 21 days in length. There are two parts to this study. A dose-escalation phase (Part I) will be used to evaluate the safety and tolerability and dose limiting toxicities, and to establish the maximum tolerated dose (MTR)/optimum biological dose (OBD) of RO6870810 when given as monotherapy or in combination with daratumumab. A dose-expansion phase (Part II) will further characterize the safety, tolerability and activity of RO6870810 as monotherapy or in combination with daratumumab at the defined expansion dose-levels.

ELIGIBILITY:
Inclusion Criteria:

* Performance status </=2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Life expectancy > 3 months
* Relapsed or refractory multiple myeloma. Participants with primary refractory myeloma only allowed in dose-escalation phase of the study.
* Prior treatment: Treated with at least three prior lines of multiple myeloma therapy including a proteasome inhibitor and an immuno modulatory agent or who are double refractory to a proteasome inhibitor and an immuno modulatory agent. Prior anti-CD38 antibody (e.g., daratumumab, isatuximab) treatment is acceptable only for participants receiving monotherapy treatment.
* Prior treatment: Treated with two or more lines of prior therapy, with disease refractory to both a proteasome inhibitor and an immunomodulatory agent, and disease progression (as defined by International Myeloma Working Group (IMWG) criteria) following treatment with an anti-CD38 monoclonal antibody given as monotherapy or in combination therapy. The most recent treatment regimen must have contained an anti-CD38 monoclonal antibody.
* Treatment with prior autologous transplant is permitted
* Documented diagnosis of symptomatic multiple myeloma, as defined by the IMWG
* Measurable disease defined as at least one of the following: serum M-protein >/=1 grams/deciliter (g/dL), urine M-protein >/= 200 milligrams/24 hours (mg/24h), serum free light chain (SFLC) assay: involved SFLCs >/= 10 mg/dL (>/= 100 mg/L) and an abnormal SFLC ratio (<0.26 or >1.65).
* Female participants of childbearing potential must have a negative serum pregnancy test within the 7 days prior to the first study drug administration.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 2 months after the last dose of RO6870810 as monotherapy, or for at least 3 months after the last dose of daratumumab.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 4 months after the last dose of RO6870810 as monotherapy, or for at least 3 months after the last dose of daratumumab.

Exclusion Criteria:

* Plasma cell leukemia defined as peripheral plasma cell count > 2000/cubic millimeter (mm^3)
* For expansion cohorts only: Primary refractory multiple myeloma defined as disease that is non-responsive in participants who have never achieved a minimal response or better with any therapy
* History of other malignancy within 2 years prior to screening, except for ductal carcinoma in situ not requiring chemotherapy, appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, low-grade, localized prostate cancer (Gleason score </= 7) not requiring treatment or appropriately treated Stage I uterine cancer
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes)
* Current or prior disease or treatment that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor
* Pregnant or breastfeeding female.
* Consumption of agents which strongly inhibit CYP3A4 enzyme, within 7 days prior to the first dose of study treatment and during the study.
* Consumption of agents which strongly induce CYP3A4 enzyme, within 14 days prior to the first dose of study treatment and during the study.
* Surgery within 21 days prior to study entry.
* Prior treatment with small molecule BET family inhibitor or receiving steroids >the equivalent of 10mg prednisone daily
* participants who are currently receiving any other investigational agent or have received an investigational agent within 30 days or 5 half-lives, whichever is longer, prior to study entry
* Uncontrolled cancer pain
* Prior anti-cancer therapy (chemotherapy, targeted agents, radiotherapy, and immunotherapy) within 14 days except for alkylating agents (e.g., melphalan) within 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Dose-Limiting Toxicities (DLTs) | From first drug administration to end of dose-escalation phase (up to approximately 1 year)
  DLTs are defined as the toxicities known and expected of RO6870810 and daratumumab that occur during a DLT assessment window of 21 days from the first administration of RO6870810 or study combination treatments, and are considered by the Investigator to be related to study treatment. DLTs are defined at specific severity levels for each term and include, but are not limited to the following Common Terminology Criteria for Adverse Events (CTCAE) terms: neutropenia, febrile neutropenia, thrombocytopenia, anemia and injection site reaction.
Objective Response Rate (ORR) | From baseline to end of study (up to approximately 2.5 years)
  ORR is defined as the percentage of participants whose confirmed best overall response is either complete response (CR, including stringent complete response [sCR]) or partial response (PR, including very good partial response [VGPR]), assessed with use of the IMWG criteria. CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow aspirates. sCR: CR plus normal free light chain (FLC) ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence. PR: >/=50% reduction of serum M-protein plus reduction in 24h urinary M-protein by >/=90% or to <200 mg/24h. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis; or >/=90% reduction in serum M-protein plus urine M-protein level <100 mg/24h. ORR= CR + sCR + PR + VGPR
Progression Free Survival (PFS) | From baseline to end of study (up to approximately 2.5 years)
  PFS is defined as the time from first study treatment to the first occurrence of disease progression (per IMWG criteria) or death, whichever occurs first. Disease progression is defined as an increase of >/= 25% from lowest response value in any one or more of the following: serum M-component, urine M-component, in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (the absolute increase must be >10 mg/dL), bone marrow plasma cell percentage (absolute level >/= 10%), definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas, development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder.
Duration of Response (DoR) | From baseline to end of study (up to approximately 2.5 years)
  DoR is defined as the time from the first occurrence of a documented objective response (sCR, CR, VGPR, or PR) to the time of first disease progression per IMWG criteria or death from any cause, whichever occurs first. Disease progression is defined as an increase of >/= 25% from lowest response value in any one or more of the following: serum M-component, urine M-component, in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (the absolute increase must be >10 mg/dL), bone marrow plasma cell percentage (absolute level >/= 10%), definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas, development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder.
Overall survival (OS) | From baseline to end of study (up to approximately 2.5 years)
  OS is defined as the time from study enrollment until death from any cause.

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | From baseline to end of study (up to approximately 2.5 years)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Maximum Observed Plasma Concentration (Cmax) of RO6870810 | Cycle 1, Days 1 and 15: predose, 0.25 hours (h), 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 24 h, 48 h; Cycle 1, Day 8 predose; all subsequent cycles predose on Day 1 and at end of treatment (EOT- up to approximately 2.5 years)
  Maximum observed concentration of RO6870810 as determined by measuring drug concentration in blood samples over time.
Time to Reach Maximum Observed Plasma Concentration (tmax) of RO6870810 | Cycle 1, Days 1 and 15: predose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 24 h, 48 h; Cycle 1, Day 8 predose; all subsequent cycles predose on Day 1 and at end of treatment (EOT - up to approximately 2.5 years)
  Time from dose administration to observed maximum serum concentration for RO6870810 as determined by measuring drug concentration in blood samples over time.
Apparent Plasma Clearance (CL/F) of RO6870810 | Cycle 1, Days 1 and 15: predose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 24 h, 48 h; Cycle 1, Day 8 predose; all subsequent cycles predose on Day 1 and at end of treatment (EOT - up to approximately 2.5 years)
  Apparent clearance (CL/F) of RO6870810, where CL is clearance and F is bioavailability (relative amount of extravascularly-administered drug that reaches systemic circulation unchanged). Determined by measuring drug concentration in blood samples over time.
Apparent Volume of Distribution (V/F) of RO6870810 | Cycle 1, Days 1 and 15: predose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 24 h, 48 h; Cycle 1, Day 8 predose; all subsequent cycles predose on Day 1 and at end of treatment (EOT - up to approximately 2.5 years)
  Apparent volume of distribution (V/F) for RO6870810, where V is the volume of distribution and F is bioavailability (relative amount of extravascularly-administered drug that reaches systemic circulation unchanged). Determined by measuring drug concentration in blood samples over time.
Area Under the Plasma Concentration-Time Curve (AUC) of RO6870810 | Cycle 1, Days 1 and 15: predose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 24 h, 48 h; Cycle 1, Day 8 predose; all subsequent cycles predose on Day 1 and at end of treatment (EOT - up to approximately 2.5 years)
  AUC for RO6870810 describes the extent of absorption from time of dose administration to time of sampling as determined by measuring drug concentration in blood samples over time.
Half-life (t1/2) of RO6870810 | Cycle 1, Days 1 and 15: predose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 24 h, 48 h; Cycle 1, Day 8 predose; all subsequent cycles predose on Day 1 and at end of treatment (EOT - up to approximately 2.5 years)
  Half-life of RO6870810 is the time elapsed for the drug concentration to decrease by half as determined by measuring drug concentration in blood samples over time.
Renal Clearance (CLr) of RO6870810 | Cycle 1, Day 1: predose, 0-1 h, 1-4 h, 4-8 h; Cycle 1, Day 15: predose, 0 h, 2 h, 6 h
  Clearance of RO6870810 through the kidneys as determined by measuring drug concentration in urine samples over time.
M-Protein Levels | At baseline, end of study (up to approximately 2.5 years)
  M-protein levels pre- and post-treatment will be monitored as a measure of biological response.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (8):
  - City of Hope, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Emory Uni - Winship Cancer Center; Hematology/Oncology, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mount Sinai - PRIME; Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Clin Rsch Institute, Durham, North Carolina
- Australia (2):
  - Scientia Clinical Research Limited, Randwick, New South Wales
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- United Kingdom (2):
  - University College London Hospitals; Clinical Research Facility, London
  - Oxford University Hospitals NHS Trust; Churchill Hospital, Oxford